CLINICAL TRIAL: NCT01344265
Title: The Correlation Between BNP and Global End Diastolic Volume
Brief Title: The Correlation Between B-type Natriuretic Peptide (BNP) and Global End Diastolic Volume
Status: Completed | Type: Observational
Sponsor: Jinhua Central Hospital (Other)
Responsible Party: Principal Investigator, Zhongheng Zhang, Dr., Jinhua Central Hospital
Other Study IDs: zh_zhang1984
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2012-09

CONDITIONS: Critically Ill
Keywords: B-type natriuretic peptide; global end diastolic volume
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- consecutive patients: there is only one group in our study

SUMMARY:
The investigators hypothesized that the serum B-type Natriuretic Peptide (BNP) level may be correlated with global end diastolic volume (GEDV) as measured by transpulmonary thermodilution technique (PiCCO). The rationale is that some animal studies have proven that BNP is released from ventricular myocardium in response to physical expansion. Such physical expansion can be measured by GEDV. If the hypothesis can be confirmed with our study, the serum level BNP can be used to monitor volume status of critically ill patient, instead of the invasive monitoring system.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients who required hemodynamic monitoring using PiCCO

Exclusion Criteria:

* patients with renal dysfunction
* those older than 80 years
* pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients who required hemodynamic monitoring using PiCCO
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
global end diastolic volume | within 12 h after measurement of BNP
  this is measured by transpulmonary thermodilution technique

CONTACTS AND LOCATIONS:
Overall Officials: Zhongheng Zhang, MD, Study Chair — Jinhua Central Hospital
Locations (1):
- Jinhua central hospital, Jinhua, Zhejiang, China